CLINICAL TRIAL: NCT04561921
Title: Effect of Magnesium Sulphate Added to Mepivacaine Hydrochloride on Inferior Alveolar Nerve Block Success in Patients With Symptomatic Irreversible Pulpitis in Mandibular Molars: A Randomized Clinical Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Ibrahim Ibrahim Ghazy Mekhimar, Resident at faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENDO 3-7-1(18/9/20)
Record Dates: First submitted 2020-09-20; First posted 2020-09-24 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Success of Inferior Alveolar Nerve Block
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- megnesium sulphate (Experimental): Injection of 1.8 mL of an anaesthetic solution containing 1% magnesium sulphate , and 1.8% mepivacaine HCL with .06mg Levonordefrin HCl during inferior alveolar nerve block.
  Interventions: Drug: Magnesium sulfate
- mepivacaine HCl (Active Comparator): Injection of 1.8 mL of a local anaesthetic solution containing 1.8% mepivacaine HCL with .06mg Levonordefrin HCL during inferior alveolar nerve block
  Interventions: Drug: Mepivacaine-Levonordefrin Hydrochloride

INTERVENTIONS:
Drug: Magnesium sulfate — patients will be given an IANB injection by adding 0.18 mL of 10% magnesium sulphate to 1.8 ml of 2% mepivacaine HCL with Levonordefrin HCl 1:20000/ 1.8 ml , after withdrawal of 0.18ml from the local anesthetic carpule by using a 100 IU insulin syringe
  Other Names: magnisol
  Arms: megnesium sulphate
Drug: Mepivacaine-Levonordefrin Hydrochloride — patients will be given an IANB injection by adding 0.18 mL of sterile distilled water to 1.8 ml of 2% mepivacaine HCL with Levonordefrin HCl 1:20000/ 1.8 ml , after withdrawal of 0.18ml from the local anesthetic carpule by using a 100 IU insulin syringe
  Other Names: Mepecaine - L
  Arms: mepivacaine HCl

SUMMARY:
the study is conducted to assess the effect of adding magnesium sulphate to mepivacaine HCl compared to mepivacaine HCl alone on the success of inferior alveolar nerve block in patients with symptomatic irreversible pulpitis in mandibular molars

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-55 years old.
2. Systemically healthy patient (ASA I or II).
3. Mandibular molar teeth with:

   * Preoperative sharp pain.
   * No widening in the periodontal ligament (PDL).
   * Vital response of pulp tissue to cold pulp tester (ethyl chloride spray)1.
   * Fully formed roots.
4. Positive patient's acceptance for participation in the study.

Exclusion Criteria:

1. Patients who had used any type of analgesic medication during the preceding 12 hours before the treatment.
2. Pregnant or nursing females.
3. Patients having significant systemic disorder (ASA III or IV).
4. Drug abusers and subjects who were on antidepressant medication.
5. Re-treatment cases.
6. Patients with a contraindication for the use of magnesium sulphate or those known to be allergic to any of the study medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-10-22 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
success of inferior alveolar nerve block measured using a numerical rating scale (NRS) | 15 minutes after injection
  Intensity of pain 15 minutes after injection during access cavity and initial file placement is recorded by the patient using a numerical rating scale(where 0= no pain ,1-3 =mild pain ,4-6= moderate pain and 7-9= severe pain )

IPD SHARING:
Plan to Share IPD: Undecided